CLINICAL TRIAL: NCT00130182
Title: A Double-Blind, Randomized, Placebo-Controlled, 28-Day Study of Denufosol Tetrasodium (INS37217) Inhalation Solution in Pediatric Patients With Cystic Fibrosis Lung Disease
Brief Title: A Study in Pediatric Patients With Cystic Fibrosis Lung Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-107
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Cystic Fibrosis
Keywords: lung disease
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases | interventions — denufosol tetrasodium

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217)

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of two dose strengths of study drug compared to placebo in pediatric patients with cystic fibrosis (CF).

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of CF
* Have an FEV1 greater than or equal to 60%
* Have oxygen saturation greater than or equal to 90% on room air
* Be clinically stable for at least 4 weeks prior to screening
* Be able to reproducibly perform spirometry maneuvers

Exclusion Criteria:

* Have clinically significant comorbidities
* Have changed their physiotherapy technique or schedule within 7 days prior to screening
* Using prior and concurrent medications according to protocol

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2005-08; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
respiratory function

SECONDARY OUTCOMES:
adverse events
change in standard safety parameters
pulmonary exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - The Children's Hospital, Denver, Colorado
  - General Clinic Research Center University of Minnesota, Minneapolis, Minnesota
  - The Minnesota CF Center, Minneapolis, Minnesota